CLINICAL TRIAL: NCT03106675
Title: MR Imaging- Guided High Intensity Focused Ultrasound (HIFU) Therapy of Bone Metastases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 133/2016
Record Dates: First submitted 2017-03-08; First posted 2017-04-10 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Bone Metastases; Bone Neoplasm; Bone Cancer; Bone Lesion
Keywords: HIFU; MR-HIFU; MRgFUs; MRI-intervention; Palliation
MeSH Terms: conditions — Bone Neoplasms

STUDY DESIGN:
Intervention Model Description: Potential participants are recruited by oncologist from oncology outpatient clinic. Pretreatment imaging with computer tomography and magnetic resonance imaging is performed to evaluate whether the patient is eligible for HIFU-treatment. Those eligible will continue to the treatment and unsuitable participants will continue in the study as a control group receiving radiation therapy.
  Participants in these groups will have follow-up MRI:s, ct:s, laboratory exams and fill in VAS (visual analog scale) and health questionnaire SF-36 regularly. Also intake of pain medication will be followed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIFU-treatment (Experimental): * Pre-treatment imaging
  * Pre-treatment questionnaires and laboratory blood samples
  * Intervention (Thermal ablation of bone metastasis with MR-HIFU device Philips Sonalleve coupled with Philips Ingenia 3.0T)
  * Follow-up (imaging, questionnaires, laboratory)
  * Follow-up pain medication usage
  Interventions: Device: Thermal ablation of bone metastasis with MR-HIFU device Philips Sonalleve coupled with Philips Ingenia 3.0T
- Radiation therapy (Active Comparator): * Pre-treatment imaging
  * Pre-treatment questionnaires and laboratory blood samples
  * Intervention (Varian Truebeam Radiotherapy System)
  * Follow-up (imaging, questionnaires, laboratory)
  * Follow-up pain medication usage
  Interventions: Device: Varian Truebeam Radiotherapy System

INTERVENTIONS:
Device: Thermal ablation of bone metastasis with MR-HIFU device Philips Sonalleve coupled with Philips Ingenia 3.0T — Procedure is performed under proper analgesia (general or local anesthesia). The intervention can be performed in areas accessible with ultrasound with no critical structures (nerves, vasculature, bowels) in proximity. Limbs and pelvis are most usually accepted locations.
  Patient is adjusted on top of the HIFU-transducer connected to MRI. First a MR-scan is performed and the treatment procedure is planned on consol. Then under MRI-guidance a point by point ablation of the target tumor is performed. During the treatment a real-time thermometry is obtained in order to avoid unwanted heating of related structures and to observe sufficient effect on treatment zone. After treatment MR-scan with gadolinium is performed to evaluate the size of ablated area.
  Other Names: Sonalleve product number 781360.
  Arms: HIFU-treatment
Device: Varian Truebeam Radiotherapy System — Conventional radiotherapy focused on bone tumor. Pretreatment planning images acquired with computer tomography
  Arms: Radiation therapy

SUMMARY:
Bone metastasis give rise to major complications that lead to significant morbidity and impairment of life quality. The most common primary for bone metastasis is prostate, lung and breast carcinoma. These three have the highest cancer incidence in the USA with up to 85% prevalence of bone metastases at the time of death. Pain from these osseous lesions can be related to mechanical or chemical factors. Pressure effects on the periosteum or adjacent neural structures can cause local or radiating pain. Hemorrhage from local bone osteolysis by osteoclastic activity causes a local release of bradykinin, prostaglandins, histamine and substance P that can irritate the endosteal nerves as well as local nerves.

The life expectancy of patients with osseous metastatic disease is variable but can be substantially longer for patients with multiple myeloma, breast or prostate cancer. Therefore, finding an effective local therapy that can improve patient quality of life and can be done at a single outpatient sitting would be beneficial.

The current and emerging treatments for osseous metastases may be considered in several categories: radiotherapy, systemic chemotherapy (cytotoxic, hormonal and radionuclides), surgical stabilization and percutaneous tumor ablation. These treatments may be applied in isolation but also frequently in combination.

MRI Guided High Intensity Focused Ultrasound (HIFU) is a completely non-invasive technology for thermal ablation. HIFU is capable of concentrating ultrasonic pressure waves to a specified region without any physical penetration of the body. The converging ultrasonic pressure wave is converted to thermal energy at the specific depth, resulting in local heating at the focus. Temperature elevation is proportional to the proton resonance frequency shift, therefore MR imaging provides accurate technique for target definition and energy deposition control. MRI guided Focused Ultrasound therapy is being performed in treatment of uterine leiomyomas (fibroids). Recently the method has gained both AMAR authorization and FDA approval, and CE approval for that indication.

Clinical trials of HIFU in bone metastases have indicated that the method is safe and gives an effective reduction of patient pain. The short- and long-term effects on tumor volume and morphology do not seem to have been evaluated thus far.

The primary objective of this trial is to evaluate effectiveness of MRI guided HIFU in the treatment of metastatic bone tumors

DETAILED DESCRIPTION:
Clinical Background

Bone metastasis give rise to major complications that lead to significant morbidity and impairment of life quality. The most common primary for bone metastasis is prostate, lung and breast carcinoma. These three have the highest cancer incidence in the USA with up to 85% prevalence of bone metastases at the time of death. Pain from these osseous lesions can be related to mechanical or chemical factors. Pressure effects on the periosteum or adjacent neural structures can cause local or radiating pain. Hemorrhage from local bone osteolysis by osteoclastic activity causes a local release of bradykinin, prostaglandins, histamine and substance P that can irritate the endosteal nerves as well as local nerves.

The life expectancy of patients with osseous metastatic disease is variable but can be substantially longer for patients with multiple myeloma, breast or prostate cancer. Therefore, finding an effective local therapy that can improve patient quality of life and can be done at a single outpatient sitting would be beneficial.

Current Treatment of Bone Metastases

The current and emerging treatments for osseous metastases may be considered in several categories: radiotherapy, systemic chemotherapy (cytotoxic, hormonal and radionuclides), surgical stabilization and percutaneous tumor ablation. These treatments may be applied in isolation but also frequently in combination.

External beam radiation therapy (EBRT) is one of the main treatments for osseous metastases. Radiation therapy creates its effect by destroying of the local tumor and inflammatory cells that are responsible for causing pain. Although the effect of radiotherapy to palliate pain and to control osseous metastatic disease is well established., there is significant relapse rate within patients who survived at least 12 weeks. Also the pain relief is often suboptimal leading to supplemental and persisting medication. Thus, the "net pain relief" less than the goal of pain relief for the total duration of life after treatment. Also, there is a limit on how much radiation can be given, this constitutes a problem in clinical oncology care.

Chemotherapy has a variable effect on bone metastases related to a number of neoplasm, drug and patient related factors. Newer systemic treatments with radionuclides and bisphosphanates have shown some success. More recently, the development of recombinant osteoprotegerin and an anti-parathyroid hormone-related protein monoclonal antibody represent promising new options for the treatment of patients with bone metastases. However, there are numbers of important factors to consider such as potential side effects of treatment and unanswered questions regarding the optimal use of systemic agents: when should treatment begin, how long must treatment be continued, and what are the optimal dose and schedule to achieve clinically meaningful anti-tumor effects?

Surgical therapy is essential in certain instances where mechanical strengthening is necessary such as an impending or occurred pathological fracture but it has little role in palliative therapy due to invasiveness and potential complications associated. Therefore, a more effective modality of local treatment for bone metastases could substantially improve quality of life.

More recently, percutaneous procedures for local tumor ablation such as radiofrequency ablation and cryotherapy have shown promise in the treatment of metastatic bone lesions.

MRI Guided High Intensity Focused Ultrasound (HIFU) is a completely non-invasive technology for thermal ablation. HIFU is capable of concentrating ultrasonic pressure waves to a specified region without any physical penetration of the body. The converging ultrasonic pressure wave is converted to thermal energy at the specific depth, resulting in local heating at the focus. Temperature elevation is proportional to the proton resonance frequency shift, therefore MR imaging provides accurate technique for target definition and energy deposition control. MRI guided Focused Ultrasound therapy is being performed in treatment of uterine leiomyomas (fibroids). Recently the method has gained both AMAR authorization and FDA approval, and CE approval for that indication.

Technical background: MR-guided intervention

Since the first report of MR-guided biopsy in 1986 there has been an increasing interest in MR-guided interventions. Technical barriers, such as the inaccessibility to the patient during imaging and the lack of MR-compatible instruments (needles, scissors, etc.) have largely been solved. Today the majority of MR-guided interventions are made in conventional closed-bore scanners alongside diagnostic imaging. Also, MRI guidance is a cost effective approach to perform these minimally invasive procedures and can in many cases replace the more invasive and in-patient based procedures.

New Possibilities: integration of MR imaging with therapy Until recently, control of destructive energy deposition has been an unresolved problem in tumor treatment. One of the greatest potentials of MRI is in monitoring the delivery of various destructive energies. Thermal monitoring is a particularly important application of interventional MRI. Thermal ablation techniques require not only good localization and targeting but also quantitative spatiotemporal control of energy deposition, which in turn requires monitoring of the thermal changes and the resulting tissue alterations.

Hyperthermia is based on slight temperature elevation (about 41° C), which requires relatively long homogenous thermal treatment of solid tumors. The main assumption of hyperthermia is that malignant cells have a higher sensitivity to thermal damage than normal ones. The temperature sensitivity of various MRI parameters (T1, diffusion, and chemical shift) can be exploited for detecting temperature changes within the critical temperature range. Compared with hyperthermia, thermal surgery uses temperatures above 55-60° C, but for a short period only.

Above 55-60 °C, proteins are denatured, and the resulting thermal coagulation causes irreversible tissue damage. Appropriate MRI sequences can demonstrate the normal margins surrounding thermal lesions, where the temperature elevation is still too low to cause cell necrosis, and, most importantly, can differentiate tissue phase transitions.

Since MRI enables monitoring, new possibilities have emerged for interstitial laser therapy, cryo- or RF-ablation and high-intensity focused ultra¬sound treatment of different tumors.

High-Intensity Focused Ultrasound (HIFU) The ability of the ultrasound imaging modality for guidance of minimally invasive procedures has been shown in various disorders but moreover, it has a significant potential to produce coagulation necrosis in exposed tissue by high-power focused sonication. By focusing high-power ultrasound beams at a distance from the source, total necrosis of tissues lying within the focal volume can be achieved without damage to the structures elsewhere in the path of the beam.

Since diagnostic ultrasound images are not sensitive enough to guide focused ultrasound thermal therapy, MRI has been used to guide this intervention. MRI thermometry based on temperature-dependent proton resonance frequency has been shown to accurately reflect thermal changes in tissue. Currently, two types of HIFU-methods are clinically used: point-by-point ablation and volumetric ablation, the latter considered more energy-efficient.

Clinical trials of HIFU in bone metastases have indicated that the method is safe and gives an effective reduction of patient pain. The short- and long-term effects on tumor volume and morphology do not seem to have been evaluated thus far.

Objectives of the study

MRI guided HIFU has been utilized to effect in treating metastatic and bening bone tumors. However detailed information upon treatment effect to pain, to the tumor volume and to the systemic immunological processes are lacking, and there are no prospective studies upon these issues. Furthermore, there is no randomized study comparing HIFU therapy to radiation therapy. There is no data upon HIFU therapy planning utilizing therapy planning software.

The primary objective of this trial is to evaluate effectiveness of MRI guided HIFU in the treatment of metastatic bone tumors:

* Safety: To further evaluate incidence and severity of adverse events associated with MRI-HIFU therapy using novel cooled technique.
* Effectiveness: To determine the effect of MRI-HIFU treatments of metastatic bone tumors. Efficacy will be determined by the level of pain relief (as measured by the Visual Analog Scale; VAS), decrease in analgesics/opiate and improved quality of life (as measured by SF36 questionnaire, in Finnish) from baseline up to 24-Weeks post HIFU treatment.

This study is designed as a prospective, two arm, nonrandomized study (Where one arm will consist of HIFU group and the other from RT group). Later on a wider randomized two arm study comparing outcomes between HIFU and RT could be executed. Furthermore, this study follows the "International Bone Metastases Consensus Working Party" on endpoint measurement for future clinical trials that was established in 2012 in conjunction with the American Society for Therapeutic Radiology and Oncology (ASTRO), the European Society for Therapeutic Radiology and Oncology (ESTRO), and the Canadian Association of Radiation Oncology (CARO)( Int J Radiat Oncol Biol Phys. 2012 Apr 1;82(5):1730-7. doi: 10.1016/j.ijrobp.2011.02.008. Epub 2011 Apr 12.)

Specific Objectives:

1. Pain relief. The change in the patient pain relief will be assessed with the Visual Analog Scale (VAS), whereas the treated patient quality of life will be assessed the quality of life questionnaire. These assessments will be performed at baseline, on treatment day, and at each follow up time point.
2. Additional data regarding dosage and frequency of analgesic consumption for the management of the metastatic bone tumor induced pain will also be collected.
3. Effect on systemic immunological processes, such as tumor markers and cytokines will be monitored via repeated blood samples.
4. Relative Safety will be evaluated using a common description of Significant Clinical Complications for patients treated in this study. This study will be performed on either the 1.5T or 3T MR scanners.
5. Temporal effect of HIFU to tissue as observed with longitudinal imaging.

The ultimate goal of this project is to establish a multidisciplinary mini-invasive environment using a 3 T MR imager with integrated high-intensity focused ultrasound.

Eventually, during the years to come, the goal is to develop and clinically validate the MR-guided HIFU-interventions and place the potential treatment option in a clinical perspective, i.e. with regard to cost, morbidity rate and outcome in following disorders

* metastatic bone disease
* cortical and intra-articular osteoid osteomas
* solitary aggressive (giant cell tumor) or malignant (plasmacytoma) lesions

Patient selection and pre -and postoperative imaging In this first phase, we include patients with intractable pain despite proper analgesics and radiotherapy treatment. These patients should not have more than three bone metastasis planned for treatment, and the source of pain should unambiguously localize to the metastasis that is considered to be sonicated. As this is a preliminary study, the anatomic location should be relatively easily accessible, i.e. the metastases should be located in the pelvic region, shoulders or in the extremities. Exclusion criteria include disease diffusely spread to bones, and the source of pain is not localized to the metastasis. Also, close proximity of a major nerve or artery is considered exclusion criteria. Other contraindications include ASA-class greater than II, when anesthesia during the procedure is required, allergy to MRI contrast medium or anesthetic agents.

MRI unit, HIFU-system and sonication. As a novel image guided therapy platform for a 3-T scanner (Ingenia, Philips Healthcare, Best, The Netherlands) we will utilize completely non-invasive MRI guided High Intensity Focused Ultrasound platform (Sonalleve, Philips Healthcare, Vantaa, Finland) to perform and study the treatment. The high intensity focused ultrasound (HIFU) tabletop harbors a 256- element phased array HIFU transducer (focal length of 140 mm, operating at 1.2 MHz). The system has different ellipsoidal treatment volumes with cross-sectional diameter from 2 to 12 mm.

The patient preparation includes preferably concise sedation e.g. with phentanyl and midazolam. However, the optimal pain relief is always individual, and is based on mutual agreement by the patient and the anesthesiologist specialized in pain relief.

After pre-sonication MR imaging, the targeted volume is defined by the radiologist, and the thermal effect is assessed by the vendor provided pulse-sequences (fast-field echo with echo planar imaging) that enable the proton resonance frequency shift (PRFS) MR thermometry method. The temperature should reach more than 55 degrees for each volume in order to achieve thermal coagulation that causes irreversible tissue damage.

Current status of the work The magnet and sonication instrumentation has been installed in early 2016, and currently the MRI is used for clinical examinations and for HIFU therapy of uterine myomas (fibroids).

Clinical significance MRI guided high-intensity focused ultrasound has the potential to become a cost-saving clinical application of MR as it integrates imaging with therapy. Lack of ionizing radiation, improved target visualization with reduced risk of injury, and have a direct impact on patient care, eventually leading to improved quality of life.

Institutional environment and resources South West Finland Imaging centre is the diagnostic hub of Turku University hospital with 60 academic radiologists and supporting staff. Department of Oncology has extensive experience in oncological research and related imaging. The team headed by Docent Roberto Blanco Sequeiros has access to the scanning facilities that will be used in the project. South West Finland Imaging centre will provide the software development tools and computers required for the project. In addition, Prof. Heikki Minn, director of department of oncology is the main collaborator and Co-PI in the research. This will facilitate adequate patient selection and monitoring of research subjects. Close collaboration will be performed with Karolinska institutet where similar project is underway with the leadership of Professor Seppo Koskinen.

Ethical Considerations Corresponding ethical approval for the proposed clinical studies has been obtained from the ethical committee at Turku University Hospital, Turku. Clinical studies will start only after organizational permit is gained. Relevant patient information will be anonymized and protected in separate electronical storage which will be protected with encryption and researcher specific login data.

Funding The project has initial funding from the EVO-funding. Additional funding has been applied from the Swedish ALF- 2017 funding (Anslag forskning, utveckling och utbildning)

ELIGIBILITY:
Inclusion criteria

* Bone metastasis
* Maximum three metastasis to be treated
* Pain that clearly locates to certain metastatic lesion
* Intolerable pain regardless of radiotherapy and adequate pain medication

Exclusion criteria from HIFU-treatment group

* ASA-group III or higher or anesthesia during procedure is required
* Metastasis not safely reachable with HIFU

Exclusion criteria from the study

- Diffusely spread metastasis on bone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-05-15 (Estimated); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in subjective pain relieve | 6 months
  Change in Visual analog scale pretreatment vs follow-up

SECONDARY OUTCOMES:
Change in tumor morphology in imaging | 6 months
  Changes in tumor features pretreatment vs follow-up (signs of progression or regression)
Change in pain medication usage | 6 months
  Change in the use of strong opiate-based pain medication intake pretreatment vs follow-up
Change in general subjective health | 6 months
  Change in SF-36 questionnaire pretreatment vs follow-up. SF36 is translated in finnish. It measures several variables related to quality of life ( eg mood, need of help)
Change in cytokine-levels | 1 month
  Change in serum inflammatory cytokines pretreatment vs follow-up
Change in tumor-specific markers | 1 month
  Change in serum tumor-specific markers (eg. PSA for prostate cancer patients) pretreatment vs follow-up

OTHER OUTCOMES:
Adverse effects | 6 months
  Possible adverse effects found during treatment or in follow up will be collected and reported

CONTACTS AND LOCATIONS:
Overall Officials: Gaber Komar, PhD, MD, Study Director — TYKS/VSKK (Turku University Hospital / Proper Finlands Imaging center); Mira Huhtala, MD, PhD student, Principal Investigator — TYKS Oncology (Turku University Hospital); Heikki Minn, Professor, MD, Study Director — TYKS Oncology; Teija O Sainio, MSc, PhD Student, Principal Investigator — TYKS/VSKK (Turku University Hospital / Proper Finlands Imaging center)

IPD SHARING:
Plan to Share IPD: Yes
Possible collaboration in the future with Karolinska Institute, Stockholm, during later stages of the study when performing randomized experiments. Data to be shared would be MRI- and CT-data, laboratory results and health-questionnaire results.

REFERENCES:
- [Background] Nielsen OS, Munro AJ, Tannock IF. Bone metastases: pathophysiology and management policy. J Clin Oncol. 1991 Mar;9(3):509-24. doi: 10.1200/JCO.1991.9.3.509. PMID 1705581
- [Background] Mantyh P. Bone cancer pain: causes, consequences, and therapeutic opportunities. Pain. 2013 Dec;154 Suppl 1:S54-S62. doi: 10.1016/j.pain.2013.07.044. Epub 2013 Jul 31. PMID 23916671
- [Background] Mercadante S, Fulfaro F. Management of painful bone metastases. Curr Opin Oncol. 2007 Jul;19(4):308-14. doi: 10.1097/CCO.0b013e3281214400. PMID 17545792
- [Background] Twycross RG. Management of pain in skeletal metastases. Clin Orthop Relat Res. 1995 Mar;(312):187-96. PMID 7543391
- [Background] Chow E, Harris K, Fan G, Tsao M, Sze WM. Palliative radiotherapy trials for bone metastases: a systematic review. J Clin Oncol. 2007 Apr 10;25(11):1423-36. doi: 10.1200/JCO.2006.09.5281. PMID 17416863
- [Background] Chow E, Zeng L, Salvo N, Dennis K, Tsao M, Lutz S. Update on the systematic review of palliative radiotherapy trials for bone metastases. Clin Oncol (R Coll Radiol). 2012 Mar;24(2):112-24. doi: 10.1016/j.clon.2011.11.004. Epub 2011 Nov 29. PMID 22130630
- [Background] Huisman M, van den Bosch MA, Wijlemans JW, van Vulpen M, van der Linden YM, Verkooijen HM. Effectiveness of reirradiation for painful bone metastases: a systematic review and meta-analysis. Int J Radiat Oncol Biol Phys. 2012 Sep 1;84(1):8-14. doi: 10.1016/j.ijrobp.2011.10.080. Epub 2012 Jan 31. PMID 22300568
- [Background] Mueller PR, Stark DD, Simeone JF, Saini S, Butch RJ, Edelman RR, Wittenberg J, Ferrucci JT Jr. MR-guided aspiration biopsy: needle design and clinical trials. Radiology. 1986 Dec;161(3):605-9. doi: 10.1148/radiology.161.3.3786706.
- [Background] Kettenbach J, Silverman SG, Schwartz RB, Hsu L, Koskinen SK, Kikinis R, Black PM, Jolesz FA. [Design, clinical suitability and future aspects of a 0.5 T MRI special system for interventional use]. Radiologe. 1997 Oct;37(10):825-34. doi: 10.1007/s001170050289. German. PMID 9454276
- [Background] Alanen J, Keski-Nisula L, Blanco-Sequeiros R, Tervonen O. Cost comparison analysis of low-field (0.23 T) MRI- and CT-guided bone biopsies. Eur Radiol. 2004 Jan;14(1):123-8. doi: 10.1007/s00330-003-1960-2. Epub 2003 Jun 25. PMID 12827428
- [Background] Jolesz FA, Silverman SG. Interventional magnetic resonance therapy. Semin Intervent Radiol 1995;12: 20-2
- [Background] Kahn T, Bettag M, Ulrich F, Schwarzmaier HJ, Schober R, Furst G, Modder U. MRI-guided laser-induced interstitial thermotherapy of cerebral neoplasms. J Comput Assist Tomogr. 1994 Jul-Aug;18(4):519-32. doi: 10.1097/00004728-199407000-00002. PMID 8040431
- [Background] Kettenbach J, Kuroda K, Hata N, Morrison P, McDannold NJ, et al. Laserinduced thermotherapy of cerebral neoplasia under MR tomographic control. Min. Invas. Ther. Allied Technol. 1998; 7/6:589- 98
- [Background] Ascher PW, Justich E, Schrottner O. Interstitial thermotherapy of central brain tumors with the Nd:YAG laser under real-time monitoring by MRI. J Clin Laser Med Surg. 1991 Feb;9(1):79-83. doi: 10.1089/clm.1991.9.79. No abstract available. PMID 10150912
- [Background] Li C, Wu L, Song J, Liu M, Lv Y, Sequeiros RB. MR imaging-guided cryoablation of metastatic brain tumours: initial experience in six patients. Eur Radiol. 2010 Feb;20(2):404-9. doi: 10.1007/s00330-009-1554-8. Epub 2009 Aug 21. PMID 19697040
- [Background] Breen MS, Lazebnik RS, Fitzmaurice M, Nour SG, Lewin JS, Wilson DL. Radiofrequency thermal ablation: correlation of hyperacute MR lesion images with tissue response. J Magn Reson Imaging. 2004 Sep;20(3):475-86. doi: 10.1002/jmri.20143. PMID 15332256
- [Background] Elias WJ, Huss D, Voss T, Loomba J, Khaled M, Zadicario E, Frysinger RC, Sperling SA, Wylie S, Monteith SJ, Druzgal J, Shah BB, Harrison M, Wintermark M. A pilot study of focused ultrasound thalamotomy for essential tremor. N Engl J Med. 2013 Aug 15;369(7):640-8. doi: 10.1056/NEJMoa1300962. PMID 23944301
- [Background] Hynynen K, Darkazanli A, Unger E, Schenck JF. MRI-guided noninvasive ultrasound surgery. Med Phys. 1993 Jan-Feb;20(1):107-15. doi: 10.1118/1.597093. PMID 8455489
- [Background] Kuroda K, Abe K, Tsutsumi S, Ishihara Y, Suzuki Y, Sato K. Water proton magnetic resonance spectroscopic imaging. Biomed Thermol 1993;13:43 - 62.
- [Background] Hindman JC. Proton resonance shift of water in the gas and liquid states. J Chem Phys 1966;44:4582 - 92.
- [Background] Chung AH, Hynynen K, Colucci V, Oshio K, Cline HE, Jolesz FA. Optimization of spoiled gradient-echo phase imaging for in vivo localization of a focused ultrasound beam. Magn Reson Med. 1996 Nov;36(5):745-52. doi: 10.1002/mrm.1910360513. PMID 8916025
- [Background] McDannold N, Clement GT, Black P, Jolesz F, Hynynen K. Transcranial magnetic resonance imaging- guided focused ultrasound surgery of brain tumors: initial findings in 3 patients. Neurosurgery. 2010 Feb;66(2):323-32; discussion 332. doi: 10.1227/01.NEU.0000360379.95800.2F. PMID 20087132
- [Background] Kohler MO, Mougenot C, Quesson B, Enholm J, Le Bail B, Laurent C, Moonen CT, Ehnholm GJ. Volumetric HIFU ablation under 3D guidance of rapid MRI thermometry. Med Phys. 2009 Aug;36(8):3521-35. doi: 10.1118/1.3152112. PMID 19746786
- [Background] Huisman M, Lam MK, Bartels LW, Nijenhuis RJ, Moonen CT, Knuttel FM, Verkooijen HM, van Vulpen M, van den Bosch MA. Feasibility of volumetric MRI-guided high intensity focused ultrasound (MR-HIFU) for painful bone metastases. J Ther Ultrasound. 2014 Oct 10;2:16. doi: 10.1186/2050-5736-2-16. eCollection 2014. PMID 25309743
- [Background] Peters RD, Hinks RS, Henkelman RM. Ex vivo tissue-type independence in proton-resonance frequency shift MR thermometry. Magn Reson Med. 1998 Sep;40(3):454-9. doi: 10.1002/mrm.1910400316. PMID 9727949
- [Background] Ikink ME, Voogt MJ, Verkooijen HM, Lohle PN, Schweitzer KJ, Franx A, Mali WP, Bartels LW, van den Bosch MA. Mid-term clinical efficacy of a volumetric magnetic resonance-guided high-intensity focused ultrasound technique for treatment of symptomatic uterine fibroids. Eur Radiol. 2013 Nov;23(11):3054-61. doi: 10.1007/s00330-013-2915-x. Epub 2013 Jun 21. PMID 23793518